CLINICAL TRIAL: NCT00532376
Title: fMRI Investigation of Depression in Patients With Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment by invitation only
Sponsor: Weill Medical College of Cornell University (Other)
Other Study IDs: 0601008320
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Epilepsy; Depression
Keywords: epilepsy; depression; fMRI; emotion
MeSH Terms: conditions — Epilepsy; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Depression is very common in epilepsy. Depression is the strongest predictor of poor quality of life in patients with epilepsy. The biological basis for depression in epilepsy remains poorly understood. This study uses functional MRI (fMRI) to examine brain response to emotional and non-emotional stimuli in healthy control subjects and in patients with epilepsy who are either depressed or not depressed. Results from this study will contribute to a better understanding of depression in epilepsy, which may eventually inform development of better treatment modalities..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Butler, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Citigroup Biomedical Imaging Center at 516 East 72nd Street, New York, New York, United States